CLINICAL TRIAL: NCT01151475
Title: Cerebral Oxygen, Blood Flow and Ammonia Uptake in Patients With Cirrhosis and an Acute Episode of HE
Brief Title: Cerebral Oxygen, Blood Flow and Ammonia Uptake in Patients With Cirrhosis and an Acute Episode of Hepatic Encephalopathy (HE)
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 24698
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Liver Cirrhosis; Hepatic Encephalopathy
Keywords: liver cirrhosis; hepatic encephalopathy; ammonia; cerebral blood flow
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We wish to study patients with liver cirrhosis during and 2 weeks after an acute episode of liver coma (hepatic encephalopathy). By means of Positron Emission Tomography we investigate; brain blood flow, brain ammonia uptake and brain oxygen consumption. We hypothesize that blood flow an oxygen consumption is diminished and ammonia uptake increased during an acute episode of hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* patients with an acute episode of hepatic encephalopathy

Exclusion Criteria:

* previous stroke

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hepatic encephalopathy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gitte Dam, Aarhus, Denmark